CLINICAL TRIAL: NCT02682667
Title: Biospecimen Procurement for Center for Immuno-Oncology Immunotherapy Protocols
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160061; 16-C-0061
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-11-18

CONDITIONS: Multiple Myeloma; Lymphoma, Non-Hodgkin; Leukemia-Lymphoma, Adult T-Cell; Hodgkin Disease; Non-Small Cell Lung Cancer
Keywords: Apheresis Products; Immunological; Diverse Malignan; Premalignant; Protein; Natural History
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Leukemia-Lymphoma, Adult T-Cell; Hodgkin Disease; Carcinoma, Non-Small-Cell Lung; Precancerous Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Cohort 1: Patients with cancer or a premalignant condition or at risk of cancer from an immunodeficiency

SUMMARY:
Background:

Cancer has a major impact in the United States and across the world. In 2015, over 1.5 million new cases of cancer were diagnosed in the U.S. Researchers want to study samples from people with cancer or a pre-malignant condition. They hope to develop more effective treatments.

Objective:

To better understand the biology of malignancies and why certain cancers respond differently to treatment.

Eligibility:

Adults at least 18 years old with cancer or a pre-cancerous condition.

Design:

Participants will be screened with a medical history, physical exam, and blood tests. Their diagnosis will be confirmed by the NCI Laboratory of Pathology.

Participants will send tissue blocks or slides from their original tumor biopsy.

At least once, participants will have a medical history, physical exam, and blood and urine tests.

Participants may have the following tests. They may have them more than once:

Apheresis. A needle in one arm removes blood. Blood is run through a machine and the sample cells are taken out. The rest of the blood is returned by a needle in the other arm.

Bone marrow aspiration and biopsy. The hipbone will be numbed. A needle will be put into the hipbone. Bone marrow will be taken out through the needle.

Piece of cancer tissue taken by a needle and syringe.

Computed tomography (CT) scan, magnetic resonance imaging (MRI) and/or positron emission tomography (PET) scan or ultrasound to help locate their tumor. For the scans, they lie in a machine that takes pictures.

A small piece of skin removed.

Participants will be contacted by phone once a year to find out how they are doing.

DETAILED DESCRIPTION:
Background:

-Immunotherapy is a promising approach to the treatment of cancer. CIO investigators are studying immunotherapy for the treatment of diverse malignant and premalignant conditions. These studies require the collection of biospecimens for research purposes.

Objectives:

* To collect and bank blood, apheresis products, tumor, body fluids, and other biospecimens from patients with cancer or a premalignant disease or at risk of cancer from an immunodeficiency.
* To collect and bank biospecimens as directed by companion CIO immunotherapy clinical trial protocols.
* To conduct nucleic acid, protein, and immunological and biological research studies on samples collected.

Eligibility:

-Patients must be 18 years of age or older with a diagnosis of cancer or a premalignant condition or an immunodeficiency that increases the risk of being diagnosed with a cancer or premalignant condition.

Design:

* Up to 500 subjects will be enrolled.
* Patients will undergo sampling of blood, apheresis products, tumor, effusions, ascites, urine, bone marrow, serum, plasma, skin, mucosa, or other tissues for banking and laboratory studies.
* No investigational or experimental therapy will be given as part of this protocol.
* Re-enrollment will be allowed for a small number of participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosis of cancer, a premalignant/neoplastic condition or disease (such as an immunodeficiency) that increases the risk of being diagnosed with a cancer or premalignant/neoplastic condition
  2. Age >=18 years of age
  3. ECOG performance status of 0-3.

  5. Ability and willingness of subject to provide informed consent

Additional inclusion criteria pertinent only for participants undergoing apheresis

1. Hemoglobin >= 8 mg/dL and platelet count > 75 K/microL
2. Weight >= 48 kg
3. Central line in place or adequate venous access

EXCLUSION CRITERIA:

1. Active concomitant medical or psychological illnesses that may increase the risk to the subject.
2. Inability to provide informed consent
3. Pregnant or breastfeeding women

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be any person over the age of 18 with a diagnosis of cancer or a premalignant disease. Participants are selected from other NIH protocols (including screening protocols) they may be co-enrolled on and can include both inpatient and outpatient.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-04-11 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Sample Acquisition | Ongoing
  Biospecimen collection for study and understanding of disease.

SECONDARY OUTCOMES:
Associations between clinical parameters, biospecimen characteristics and patient demographics | Ongoing
  Correlation of these characteristics with disease.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Norberg, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data will be shared from the time of upload to dbGaP.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@@@@@@@Genomic IPD will be shared through dbGaP, per rules of the database, for purposes of genomic analysis.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-C-0061.html